CLINICAL TRIAL: NCT04961554
Title: Locoregional Anesthesia of the V3 and Limited Mouth Opening
Brief Title: Evolution of Mouth Opening After Mandibular Block
Acronym: OBloc
Status: Withdrawn | Type: Observational
Why Stopped: 1. Short defense deadline
  2. Activity cessation of the maxillofacial surgery department at Pitié Salpêtrière hospital
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210543
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-10

CONDITIONS: Trismus
Keywords: mandibular block; limited mouth opening; trismus; loco-regional anesthesia; pain; video laryngoscope; awake flexible fiberoptic intubation; difficult airway management; head and neck surgery; maxillofacial surgery
MeSH Terms: conditions — Trismus; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients presenting with limited mouth opening: Adult patients presenting with limited mouth opening not allowing intubation by videolaryngoscopy, on mandibular surgical pathology requiring general anesthesia.
  Interventions: Other: loco-regional anesthesia

INTERVENTIONS:
Other: loco-regional anesthesia — demonstrate that the mouth opening (measured in millimeters) of a patient treated for mandibular surgery with a very limited opening (defined by a threshold less than 20mm, not allowing the passage of a video laryngoscope blade per route buccal) is more important after locoregional anesthesia of the V3 than before anesthesia.

SUMMARY:
Trismus is an involuntary contracture of the masticatory muscles, blocking the opening of the jaw, first intermittent then permanent and irreducible. Trismus is the result of pain or spasm or even muscle fibrosis, due to infectious, inflammatory or tumoral involvement of the masticatory muscles.

During any anesthesia, control of the patient's upper airways is a major issue. Orotracheal intubation is the gold standard. Trismus will therefore complicate this management of the airways. This trismus can prevent the realization of a classic intubation, by the inability to use a laryngoscope or video laryngoscope, in favor of awake fiberoptic intubation, a technique that causes discomfort during the procedure, then a state of post-traumatic stress.

Mandibular block is increasingly used in the analgesia of mandibular surgeries thanks to the simplicity of the technique and its good efficiency. It has been described that the mandibular locoregional anesthesia made it possible to remove the trismus due to a dental infection, allowing the realization of a surgical gesture under good conditions. In addition, authors have described V3 block as a technique that could improve the safety of anesthesia in patients with acute trismus, by avoiding the need for awake nasofibroscopy intubation. One study showed that performing locoregional anesthesia of the mandibular nerve improved the mouth opening in patients with mandibular fracture. The investigators wondered if this locoregional anesthesia could also work on other types of trismus such as infectious, tumoral and osteoradionecrosis trismus.

During preoperative consultation, anesthesists usually measure the mouth opening. In our study, anesthesists will also measure the mouth opening after performing locoregional anesthesia of the V3 nerve (mandibular block). In addition to the measurement made before the start of the anesthetic treatment, research provides for three other measurements of the mouth opening using a rule (millimeters), taken at different times : after sedation, after performing locoregional anesthesia and after curarization. The investigators will also collect the cause of the limited mouth opening, the duration of development. The investigators will study pain at rest and when opening the mouth, under sedation, when performing the block, then when opening the mouth after performing the block. The presence of edema next to the area of locoregional anesthesia, the type of product used for sedation and locoregional anesthesia, the intubation technique performed, as well as the difficulty experienced by the operator will be collected

DETAILED DESCRIPTION:
The aim of this study is to avoid recourse to awake fiberoptic intubation, which causes discomfort during the procedure and post-traumatic stress disorder, in patients with a very limited mouth opening (less than 20mm) and who must undergo anesthesia general for mandibular surgery.

As a reminder, the definition of limited mouth opening (MO) is a lower 35mm mouth opening, according to the Société française d'anesthésie-réanimation (SFAR) recommendations. The investigators define a very limited mouth opening as a mouth opening that does not allow a video laryngoscope blade to be inserted into the patient's mouth (less than 20mm).

During preoperative consultation, anesthesists usually measure the mouth opening. In our study, anesthesists will also measure the mouth opening after performing locoregional anesthesia of the V3 nerve (mandibular block). In addition to the measurement made before the start of the anesthetic treatment, research provides for three other measurements of the mouth opening using a rule, taken at different times.

The management is carried out exclusively by the investigators, the latter being anesthetists. Thus, the evaluation of the different mouth openings using a ruler (in millimeters), the evaluation of the pain using the numerical scale, the administration of sedation, the realization of loco-regional anesthesia, intraoperative and postoperative anesthetic management will be carried out by one and the same person qualified in anesthesia for maxillofacial surgery.

In summary, six key steps for our study will be carried out by the anesthetist-resuscitator:

1. Initial patient assessment with assessment of pain and mouth opening (millimeters)
2. Introduction of sedation, and reassessment of pain and mouth opening (millimeters)
3. Performing a locoregional anesthesia of the V3 for analgesic purposes
4. Reassessment of pain, mouth opening (millimeters) at least 15 minutes from the block, and possibly the Mallampati score. Mallampati score is systematically noted as part of the treatment.
5. Induction of anesthesia, and reassessment of the mouth opening after curarization.
6. Assessment of the difficulty of intubation (difficulty in passing the videolaryngoscope blade, Cormack score applied to videolaryngoscopy).

The anesthetist who performs the locoregional anesthesia will collect the data using the standardized questionnaire created for the study, notifying the key clinical elements of airway management that are being research within the framework of care, according to the rules of good anesthesia practice.

These data, collected as part of the treatment, will be:

* The cause of the limited mouth opening
* The duration of development
* Pain at rest and when opening the mouth, then under sedation, when performing the block, then when opening the mouth after performing the block, using the digital scale
* The presence of edema next to the area of locoregional anesthesia of V3
* The type of product used for sedation and locoregional anesthesia
* The mouth opening (measured in millimeters using a ruler) before any gesture then after sedation, 15 minutes from the completion of the V3 nerve block, and after curarization.
* The investigators will also evaluate the evolution of the Mallampati score at the same time, as part of the treatment.
* The intubation technique performed, as well as the difficulty experienced by the operator.

These data will be pseudonymized.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient with a mouth opening defined as very limited (<20mm)
* Patient scheduled for mandibular surgery, with an indication for a V3 block for analgesic purposes
* Patient informed and not opposed to the study

Exclusion Criteria:

* Allergy to local anesthetics
* Patient under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting with a limited mouth opening that does not allow intubation by videolaryngoscopy, with mandibular surgical pathology requiring general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-02 (Estimated); Primary Completion 2024-04-02 (Estimated); Study Completion 2024-04-02 (Estimated)

PRIMARY OUTCOMES:
Measure of patient's mouth opening | during surgery
  The main outcome is the measure of patient's mouth opening (in millimeters) in the minutes preceding and following the mandibular block.
  The mouth opening will be measured using a ruler with 4 defined times:
  * Before any anesthesia
  * After sedation
  * 15min from the realization of the loco-regional anesthesia
  * After curarization, just before intubation. These different measurements will be carried out by a ruler, and by a single operator for these 4 measurements.

SECONDARY OUTCOMES:
Assessement of Etiology of limited mouth opening (osteoradionecrosis, tumor, infection) | during surgery
  Potentially predictive of the success of locoregional anesthesia on mouth opening
Mallampati score | before locoregional anesthesia
  Predictive of intubation difficulty

CONTACTS AND LOCATIONS:
Overall Officials: Claire Gourbeix, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Anesthésie-Réanimation Pôle Tête et Cou, Hôpital Pitié-Salpêtrière, Paris, France